CLINICAL TRIAL: NCT06059703
Title: Biomarkers in the Etiology of Idiopathic Intracranial Hypertension
Acronym: BEHIND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL22_0565
Record Dates: First submitted 2023-09-04; First posted 2023-09-29 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Idiopathic Intracranial Hypertension
Keywords: Idiopathic intracranial hypertension HII; Intracranial pressure elevation (ICP); Transverse venous sinus stenosis; Cerebral venous stenting; Blood biomarkers
MeSH Terms: conditions — Pseudotumor Cerebri; Intracranial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Idiopathic intracranial hypertension (IHH) patient (Experimental): IHH patient with bilateral stenosis of the transversal sinus
  Interventions: Procedure: Blood punction; Procedure: Central blood sampling; Procedure: Intracranial pressure measurement

INTERVENTIONS:
Procedure: Blood punction — Peripheral blood sampling (5 ml) at inclusion and 3 months after treatment
Procedure: Central blood sampling — Central blood sampling (2 ml) at inclusion and 3 months after treatment
Procedure: Intracranial pressure measurement — Intracranial pressure measurement at sinus level with micro-catheter at inclusion and 3 months after treatment

SUMMARY:
Idiopathic intracranial hypertension (IIH) is a condition characterized by an increase in intracranial pressure (ICP), papilledema with a risk of permanent visual loss, and severe headaches that profoundly affect quality of life.

To date the exact pathophysiology of IIH remains unknown. IIH is considered a complex neurometabolic and neuroendocrine disorder, favored by female gender, and obesity.

In the majority of patients (80% of the cases) IIH is associated with obstruction of cerebral venous drainage with stenosis of the transverse sinus. This stenosis may be the main underlying cause in the so-called "venogenic" form of IIH. Equally, in the absence of a stenosis, obstruction may occur when otherwise normal venous sinuses are compressed by the increased ICP, the so-called "non-venogenic" form of IIH. An innovative treatment of IIH with associated venous stenosis includes stenting of the transverse sinus stenosis. This strategy may allow resolution of papilledema and ICP reduction rates up to 80%.

Although the pathogenesis of IIH is still poorly understood, inflammatory mechanisms, autoimmune reactions, and hormonal abnormalities of notably androgens, have been proposed to contribute to its pathophysiology. The function of the blood-brain barrier (BBB) has been studied by determining the prevalence of extravasation of endogenous proteins such as fibrinogen.

A growing body of the literature shows a correlation between increased ICP and metabolic/hormonal changes.

The improvement of IIH treated with acetazolamide and/or stenting appears to correlate with the reduction of ICP. Yet the association of this reduction with metabolic changes at the peripheral and central blood level as well as the CSF remains unclear. The search for specific inflammatory, immunological and hormonal biomarkers in patients with IIH and their variation in relation to the ICP should provide a better understanding of its etiology.

DETAILED DESCRIPTION:
Idiopathic intracranial hypertension (IIH) is a condition characterized by increased intracranial pressure (ICP) of unknown cause, papilledema with the risk of permanent visual impairment, and severe headaches that profoundly impair quality of life, often becoming irreversible despite resolution of the IIH and disappearance of the papilledema.

IIH is diagnosed using the modified Dandy criteria,based on increased ICP (>25 cm H2O on lumbar puncture (LP) performed in the lateral decubitus), papilledema, normal cerebrospinal fluid (CSF) and brain imaging that rules out all other causes of intracranial hypertension.

IIH is attracting growing interest among clinicians as its incidence and prevalence increases. IIH predominates in women of childbearing age with increased body mass index (BMI) . In the United Kingdom its incidence has doubled in 14 years, rising from 3.5 per 100,000 to 7.69 per 100,000 in the female population between 2002 and 2016 (+ 108%)

To date, the exact pathophysiology of IIH remains unknown. IIH is considered to be a complex neurometabolic and neuroendocrine disorder favored by female gender and obesity. Hypothesized mechanisms include inflammatory, autoimmune and hormonal abnormalities, of notably androgens.

In the majority of patients (80% of the cases) IIH is associated with obstruction of cerebral venous drainage with bilateral stenosis of the transverse sinus. This stenosis may be the main underlying cause in the so-called "venogenic" form of IIH. Equally, in the absence of a stenosis, obstruction may occur when otherwise normal venous sinuses are compressed by the increased ICP, the so-called "non-venogenic" form of IIH.

The therapeutic management of IIH has a triple objective: i) to treat the underlying cause(s); ii) to protect vision, and iii) to reduce the impact of headaches. Unfortunately, current treatments (weight loss, drug therapy with acetazolamide or Diamox, and/or anti-migraine treatment) are not very effective. It has been argued to favor treatments targeted directly at the cause of the increased ICP, and therefore at its etiology. A promising innovative treatment of venogenic IIH includes stenting of the transverse sinus stenosis. It has been associated with papilledema and ICP reduction rates up to 80% .

However, venous stenosis is probably not the only underling mechanism of increased ICP. Accordingly, the role of metabolic, hormonal and inflammatory mechanisms requires further investigation. It has been found that serum levels of tumor necrosis factor-alpha (TNF-α) were significantly higher in patients with IIH compared with healthy controls . The serum TNF-α level was a significant predictor of the severity of visual field disease. Interestingly, by evaluating adipokine and cytokine levels to identify possible serum markers of inflammation in the pathophysiology of IIH, it was observed that interleukin (IL)-1β levels were significantly higher in the IIH group compared to the control group, whereas IL-8 and TNF-α levels were significantly lower. Although the latter seems in contrast with previous findings, the presence of recurrent relapses - known to enhance chronic inflammatory protective mechanisms and thus increased TNF- α levels, may explain this difference. Serum levels seem thus to be altered (IL-1β, IL-8 and TNF-α) and may be associated with the pathogenesis of IIH. Cytokines might be valuable as prognostic markers in IIH to predict possible relapse.

Given the established association between increased perivascular expression of the water channel aquaporin-4 (AQP4), degeneration of pericytes, capillary basement membranes, and blood-brain barrier (BBB) dysfunction in patients with IIH, the BBB function was investigated by determining the prevalence of extravasation of endogenous proteins such as fibrinogen. Signs of BBB dysfunction, measured by the surface area of extravasated fibrinogen/fibrin, were significantly more pronounced in IIH patients than in reference subjects and demonstrated BBB dysfunction. The increased degree of BBB dysfunction was associated with increased perivascular AQP4 immunoreactivity. AQP4 appears to play a major role in "flushing" brain parenchyma through interstitial fluid, thus also affecting inflammation-generating substances including fibrinogen extravasation.

Given the obesity of IHH patients, the involvement of leptin, a hormone associated with the sensation of hunger, was also investigated and found to be elevated. Its regulation mechanism of Na/K ATPase in the choroid plexus and CSF secretion has been postulated . It is also important to point out that between 40%-50% of women with IIH suffer from polycystic ovary syndrome, which is characterized by dysregulation of sex hormones . Finally, mineralocorticoids, such as 11β-hydroxysteroid dehydrogenase, have been studied in the pathogenesis of IIH following their potential role in the regulation of Na/K ATPase at the level of the choroid plexus .

Taken together, these studies seem to highlight a wide range of processes for which biomarkers associated with IIH are starting to emerge, but that are still poorly understood. The lack of prospective studies and the small number of patients included in most of the studies carried out so far, impedes conclusions on the role of these factors in the etiology of IIH.

Nevertheless, improvement of IIH treated with acetazolamide and/or stenting seems to correlate with a reduction in ICP, but the association of this reduction with metabolic changes in peripheral, central blood and/or CSF needs to be clarified. The identification of specific inflammatory, immunological and hormonal biomarkers in patients with IIH and their variation in relation to ICP variation should provide a better understanding of its etiology. Biomarkers related to disease severity should allow, in the longer term, proposing alternative treatments.

Advances in endovascular techniques have made it possible to measure ICP at the level of the intracerebral venous system, and to take biological samples at the central (intracerebral) level in order to identify biomarkers associated with clinical severity, and to study their variation as a function of i) normalization of intracranial pressure after treatment with stenting or Diamox, ii) changes in ophthalmological symptoms and headaches.

To date, there are very few prospective cohorts analyzing the biology of patients with IIH. This study will help in the search for biomarkers of the pathology's severity, with a dual aim: 1) to stimulate understanding of the pathophysiology of IIH, which to date remains largely unknown; 2) to develop new drug treatments targeting the mechanisms of increased ICP.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Patients with newly diagnosed untreated HII (following the modified Dandy criteria) with normal CSF composition, abnormal CSF pressure at the lumbar puncture (>25 cm H2O), and significant pressure gradient at the level of the stenosis (≥8 mmHg)
* Presence of bilateral transverse sinus stenosis (or unilateral with hypoplastic contralateral sinus).

Exclusion Criteria:

* Allergy to contrast media (nickel, titanium)
* Allergy or contraindication to antiplatelet agents
* Patient on anti-inflammatory treatment
* Chronic inflammatory disease
* History of intracranial venous thrombosis, cerebral hemorrhage, thrombophilia
* History of intracranial tumor
* Fulminant IIH with acute visual loss
* Optic nerve atrophy with papilledema (chronic IIH)
* Female being pregnant, breastfeeding, or planning to become pregnant in the next 3 months
* Major comorbidities with high procedural risk
* Life expectancy < 6 months
* Adult under guardianship or conservatorship or incapacitated
* Refusal of consent after receiving all necessary information
* Not covered by or not a beneficiary of the French social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2025-11-27 (Estimated); Study Completion 2026-03-27 (Estimated)

PRIMARY OUTCOMES:
intracranial pressure (ICP) blood biomarker correlation | Change over time before (at inclusion) and 3 months after IIH treatment (follow-up)
  The correlation (Pearson's r) between blood biomarkers and ICP measured before and after IIH treatment. Pearson's r will be calculated with a multivariate stepwise linear regression to identify those biomarkers that can explain a change in ICP. The blood biomarkers are extracted from peripheral and central venous blood. The ICP is measured at torcular level.
  The blood biomarkers include:
  * Inflammatory markers (pg/mL):
    * Osteopontin, γ&β-chain fibrinogen, α1-acid glycoprotein 2 et haptoglobin
    * Inflammatory cytokines : INFγ, IL-2, IL-10, IL-4, IL-12p70, IL-6, IL-13, IL-8, IL-1β, TNF-α, IL-17, IL-23, IGF-1, TGFβ1
    * Chemokines: Fractalkine, SDF-1, CX3CL1, MCP-1, CCL3, CCL5
  * BBB integrity markers (pg/mL): S100b, GFAP, Neurofilament light-chain, Neuronal specific enolase, Uch-L1
  * Headache associated markers (pg/mL): Calcitonin Gene Related-Peptide, Glucagon-Like Peptide
  * Hormonal markers (ng/mL): 11β-HSD1, Glucagon-like peptide-1, DHEAS, Leptin, estradiol, and testosterone

SECONDARY OUTCOMES:
Headache severity | change over time before (at inclusion) and 3 months after IIH treatment (follow-up)
  Calculation of the correlation (multivariate regression, Pearson's r) between variations in blood biomarker concentrations (inflammatory, BBB, headache and hormonal) and headache severity as determined by the HIT-6 (6-item questionnaire, scores range from 36 to 78; the higher the score, the greater the impact of headaches on quality of life.).
  The correlation will be defined:
  * The correlation before treatment
  * The correlation after treatment
  * The change over time
Body mass index (BMI) | change over time before (at inclusion) and 3 months after IIH treatment (follow-up)
  Calculation of the correlation (multivariate regression, Pearson's r) between the concentration of all blood biomarkers (inflammatory, Blood-Brain Barrier, headache and hormonal) and the Body-Mass-Index (expressed in kg/m² by combining weight and height).
  The correlation will be defined:
  * The correlation before treatment
  * The correlation after treatment
  * The change over time
Optic fibre layer (RNF) thickness | Before (at inclusion) and 3 months after treatment (follow-up)
  Calculation of the correlation (multivariate regression, Pearson's r) between the variation in concentration of all blood biomarkers (inflammatory, Blood brain barrier, headache and hormonal) and the severity of papilledema, which is quantified by the average thickness (µm) of the optic fibre layer (RNF)
  The correlation will be defined:
  * The correlation before treatment
  * The correlation after treatment
  * The change over time
Transverse sinus stenosis | change over time before (at inclusion) and 3 months after IIH treatment (follow-up)
  Quantify by means of a correlation analysis (linear regression, Pearson's r) whether changes in de degree of traverse sinus stenosis can be an indirect indication of ICP increase. Traverse sinus stenosis is measured on T2* Magnetic resonance imaging (MRI) imaging by measuring the dilation of the optic nerve sheath in mm.
Cerebral blood flow | change over time before (at inclusion) and 3 months after IIH treatment (follow-up)
  Quantify by means of a multivariate regression analysis (Pearson's r) whether cerebral blood flow characteristics are related to variations in ICP and headache severity over time. The cerebral blood flow is analyzed with arterial spin labeling MRI, the headache severity is evaluated with the HIT-6 questionary (6-item questionnaire, scores range from 36 to 78; the higher the score, the greater the impact of headaches on quality of life.).
MRI contrast enhancement | change over time before (at inclusion) and 3 months after IIH treatment (follow-up)
  Evaluate the link between MRI 3DT1 contrast enhancement after gadolinium injection and the biomarkers of blood-brain barrier integrity over time with a linear regression (Pearson's r).

CONTACTS AND LOCATIONS:
Overall Officials: Federico CAGNAZZO, MD, Study Director — University Hospital of Montpellier - Gui de Chauliac
Locations (1):
- University Hospital of Montpellier - Gui de Chauliac, Montpellier, France

REFERENCES:
- [Background] Markey KA, Mollan SP, Jensen RH, Sinclair AJ. Understanding idiopathic intracranial hypertension: mechanisms, management, and future directions. Lancet Neurol. 2016 Jan;15(1):78-91. doi: 10.1016/S1474-4422(15)00298-7. Epub 2015 Dec 8. PMID 26700907
- [Background] Mollan SP, Aguiar M, Evison F, Frew E, Sinclair AJ. The expanding burden of idiopathic intracranial hypertension. Eye (Lond). 2019 Mar;33(3):478-485. doi: 10.1038/s41433-018-0238-5. Epub 2018 Oct 24. PMID 30356129
- [Background] Riggeal BD, Bruce BB, Saindane AM, Ridha MA, Kelly LP, Newman NJ, Biousse V. Clinical course of idiopathic intracranial hypertension with transverse sinus stenosis. Neurology. 2013 Jan 15;80(3):289-95. doi: 10.1212/WNL.0b013e31827debd6. Epub 2012 Dec 26. PMID 23269597
- [Background] Toscano S, Lo Fermo S, Reggio E, Chisari CG, Patti F, Zappia M. An update on idiopathic intracranial hypertension in adults: a look at pathophysiology, diagnostic approach and management. J Neurol. 2021 Sep;268(9):3249-3268. doi: 10.1007/s00415-020-09943-9. Epub 2020 May 27. PMID 32462350
- [Background] Dhungana S, Sharrack B, Woodroofe N. Cytokines and chemokines in idiopathic intracranial hypertension. Headache. 2009 Feb;49(2):282-5. doi: 10.1111/j.1526-4610.2008.001329.x. PMID 19222599
- [Background] Zanello SB, Tadigotla V, Hurley J, Skog J, Stevens B, Calvillo E, Bershad E. Inflammatory gene expression signatures in idiopathic intracranial hypertension: possible implications in microgravity-induced ICP elevation. NPJ Microgravity. 2018 Jan 11;4:1. doi: 10.1038/s41526-017-0036-6. eCollection 2018. PMID 29354685
- [Background] Nicholson P, Brinjikji W, Radovanovic I, Hilditch CA, Tsang ACO, Krings T, Mendes Pereira V, Lenck S. Venous sinus stenting for idiopathic intracranial hypertension: a systematic review and meta-analysis. J Neurointerv Surg. 2019 Apr;11(4):380-385. doi: 10.1136/neurintsurg-2018-014172. Epub 2018 Aug 30. PMID 30166333
- [Background] Fahmy EM, Rashed LA, Mostafa RH, Ismail RS. Role of tumor necrosis factor-alpha in the pathophysiology of idiopathic intracranial hypertension. Acta Neurol Scand. 2021 Nov;144(5):509-516. doi: 10.1111/ane.13482. Epub 2021 Jun 15. PMID 34131899
- [Background] Samanci B, Samanci Y, Tuzun E, Altiokka-Uzun G, Ekizoglu E, Icoz S, Sahin E, Kucukali CI, Baykan B. Evidence for potential involvement of pro-inflammatory adipokines in the pathogenesis of idiopathic intracranial hypertension. Cephalalgia. 2017 May;37(6):525-531. doi: 10.1177/0333102416650705. Epub 2016 May 18. PMID 27193133
- [Background] Hasan-Olive MM, Hansson HA, Enger R, Nagelhus EA, Eide PK. Blood-Brain Barrier Dysfunction in Idiopathic Intracranial Hypertension. J Neuropathol Exp Neurol. 2019 Sep 1;78(9):808-818. doi: 10.1093/jnen/nlz063. PMID 31393574
- [Background] Eide PK, Eidsvaag VA, Nagelhus EA, Hansson HA. Cortical astrogliosis and increased perivascular aquaporin-4 in idiopathic intracranial hypertension. Brain Res. 2016 Aug 1;1644:161-75. doi: 10.1016/j.brainres.2016.05.024. Epub 2016 May 14. PMID 27188961
- [Background] Ball AK, Sinclair AJ, Curnow SJ, Tomlinson JW, Burdon MA, Walker EA, Stewart PM, Nightingale PG, Clarke CE, Rauz S. Elevated cerebrospinal fluid (CSF) leptin in idiopathic intracranial hypertension (IIH): evidence for hypothalamic leptin resistance? Clin Endocrinol (Oxf). 2009 Jun;70(6):863-9. doi: 10.1111/j.1365-2265.2008.03401.x. Epub 2008 Sep 2. PMID 18771566
- [Background] Markey KA, Uldall M, Botfield H, Cato LD, Miah MA, Hassan-Smith G, Jensen RH, Gonzalez AM, Sinclair AJ. Idiopathic intracranial hypertension, hormones, and 11beta-hydroxysteroid dehydrogenases. J Pain Res. 2016 Apr 19;9:223-32. doi: 10.2147/JPR.S80824. eCollection 2016. PMID 27186074